CLINICAL TRIAL: NCT03600441
Title: Open-label, Single-Arm, Phase 2 Study of Oral HDAC-inhibitor Abexinostat in Patients With Relapsed or Refractory Follicular Lymphoma (FORERUNNER)
Brief Title: Study of Abexinostat in Patients With Relapsed or Refractory Follicular Lymphoma
Acronym: FORERUNNER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xynomic Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYN-601
Record Dates: First submitted 2018-06-23; First posted 2018-07-26 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Follicular Lymphoma
Keywords: cancer
MeSH Terms: conditions — Lymphoma, Follicular; Neoplasms | interventions — abexinostat

STUDY DESIGN:
Intervention Model Description: open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abexinostat (Experimental): Abexinostat tablets will be administered orally at 80 mg (4 × 20 mg tablets) BID (twice a day) 4 hours apart for 7 days in a "one week on, one week off" schedule (on Days 1 to 7 and Days 15 to 21 of each 28-day cycle).
  Interventions: Drug: Abexinostat

INTERVENTIONS:
Drug: Abexinostat — Abexinostat tosylate salt is formulated into an oral tablet formulation and is available in 20 mg strength.

SUMMARY:
This study in patients with relapsed/refractory follicular lymphoma who have undergone at least 3 lines of therapy. Patients will receive abexinostat 80 mg (4 × 20 mg tablets) twice a day (BID) in a "one week on, one week off" schedule.

DETAILED DESCRIPTION:
Patients will be evaluated for objective response, Duration of Response (DOR), Progression Free Survival (PFS), Clinical Benefit Rate (CBR), Overall survival (OS), safety and tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and changes in health related quality of life. Patients may receive treatment until disease progression, death, unacceptable toxicity, or withdrawal of consent. An independent data safety monitoring committee (iDMC) will evaluate the data pertaining to the futility and decide whether the study should stop or continue to the second stage. If the study continues to the second stage, a total of 139 patients will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Is able to understand and voluntarily sign an informed consent document before any study related assessments/procedures are conducted.
* Has histologically confirmed Grade 1, 2, or 3a follicular lymphoma.
* Has follicular lymphoma that has relapsed after (progressed after 6 months from the start of therapy) or is refractory to the last line of therapy (no response or progression within 6 months from the start of therapy) and needs treatment (must have at least 1 lymph node or extranodal lymphoid malignancy radiologically measuring ≥ 3 cm in its longest diameter).
* Female patients must fulfil the following criteria:

  a. Be of non-childbearing potential, defined as follows: i. Postmenopausal (ie, ≥ 1 year without any menses) prior to Screening, or ii. Documented surgically sterile (≥ 1 month prior to Screening)
* Male patients must agree not to donate sperm starting from the time of Screening, throughout the study, and until after 90 days following the last dose.
* Use highly effective forms of birth control (women of childbearing potential only), which include the following:

  i. Consistent and correct use of established oral contraception ii. Established intrauterine device or intrauterine system iii. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
* Female patients must agree not to breastfeed starting from the time of Screening, throughout the study, and until after 90 days following the last dose.
* Male patients and their female spouse/partners who are of childbearing potential must use highly effective contraception methods consisting of 2 forms of birth control (at least 1 of which must be a barrier method) from the time of Screening, throughout the study, and until after 90 days following the last dose.
* Male patients must agree not to donate sperm starting from the time of Screening, throughout the study, and until after 90 days following the last dose.

Exclusion Criteria:

* Has diagnosis of Grade 3b follicular lymphoma, or transformation to diffuse large B-cell lymphoma
* Has a history of central nervous system lymphoma (either primary or secondary).
* Has had prior treatment with abexinostat.
* Has had allogeneic stem cell transplant within the last 6 months, or autologous stem cell transplant within the last 3 months before enrollment
* Has any types of cardiac impairment at the time of enrollment
* Has received any investigational medication within 30 days or 5 half-lives prior to Day 1, whichever is longer
* Has prior history of malignancies, other than follicular lymphoma, unless the patient has been free of the disease for ≥ 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2018-08-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical effect of abexinostat | Time frame up to 100 months
  Complete response (CR) or partial response (PR) according to the Lugano 2014 criteria as determined by an Independent Review Committee (IRC).

SECONDARY OUTCOMES:
Duration of response | At the end of cycle 2 (each cycle is 28 days) and through study completion, assessed up to 100 months.
  Duration of response defined as the time from first documented evidence of CR or PR until disease progression or death from any cause among patients who achieve an objective response, according to the Lugano 2014 criteria as determined by an IRC.
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  Defined as the time from the start of treatment until disease progression or death assessed using the Lugano 2014 criteria as determined by an IRC.
Clinical Benefit | At the end of cycle 2 (each cycle is 28 days) and through study completion, assessed up to 100 months.
  Defined as the best from CR, PR, or stable disease (SD) according to the Lugano 2014 criteria as determined by an IRC.
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  Defined as the time from the start of treatment until death from any cause or last contact.
Duration of response | At the end of cycle 2 (each cycle is 28 days) or from date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  Defined as the time from first documented evidence of CR or PR from any cause among patients who achieve an objective response, according to the RECIL 2017 as determined by an IRC. Duration of response will be evaluated once more using the RECIL 2017 with the inclusion of Minor Response (MR) lasting ≥ 6 months.
Incidence of adverse events | At the end of cycle 2 (each cycle is 28 days) or from date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  Safety as measured by the incidence of adverse events
Incidence of serious adverse events | At the end of cycle 2 (each cycle is 28 days) or from date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  Safety as measured by the serious of adverse events (SAE)
Incidence of non-serious adverse events | At the end of cycle 2 (each cycle is 28 days) or from date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  Safety as measured by the non-serious of adverse events
Change in the interval corrected for heart rate (QTc) interval | At the end of cycle 2 (each cycle is 28 days) or from date of randomization until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months
  Change from baseline in the QTc interval.

CONTACTS AND LOCATIONS:
Overall Officials: Connie W Batlevi, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (15):
- United States (9):
  - Advocate Medical Group - Park Ridge, Luther Lane - Oncology, Park Ridge, Illinois
  - Norton Cancer Institute - St. Matthews Campus, Louisville, Kentucky
  - Clinical Research Alliance Inc, Lake Success, New York
  - Manhattan Hematology Oncology Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Bone Marrow Transplant Hematology Oncology Associates, Pittsburgh, Pennsylvania
  - Arlington Cancer Center, Arlington, Texas
  - Central Texas Veterans Health Care System - NAVREF, Temple, Texas
  - Vista Oncology Inc. PS, Olympia, Washington
- Centre Hospitalier de Perpignan, Perpignan, Pyrénées-Orientales, France
- Spain (5):
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Guipúzcoa
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital del Mar, Barcelona
  - C.H. Regional Reina Sofia, Córdoba
  - Hospital Universitario Infanta Leonor, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FDA Safety Alerts — https://www.fda.gov/Safety/Recalls/